CLINICAL TRIAL: NCT05378464
Title: Phase 1 Study of Adoptive T Cell Therapy Following HER2-Pulsed Dendritic Cell Vaccine and Pepinemab / Trastuzumab in Patients With Metastatic HER2-Positive Breast Cancer
Brief Title: Adoptive T Cell Therapy Following HER2-Pulsed Dendritic Cell Vaccine & Pepinemab /Trastuzumab in Patients w/ Metastatic HER2+ Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Vaccinex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21378
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer
Keywords: Breast Cancer; T-Cell therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Vaccines; Trastuzumab; pepinemab; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- T-Cell therapy dose level 1 (Experimental): Participants will begin treatment with pepinemab and trastuzumab, and begin DC1 vaccines. After 6 weeks of DC1 vaccines, blood will be collected for t-cell therapy, and patients will then be treated with IL-15 Expanded HER2 specific CD4+ Th1 cell 0.5.0-2.5 x 10^8, IL-7 and Expanded HER2 specific CD4+ Th1 cell 0.5.0-2.5 x 10^8.
  Interventions: Biological: Dendritic Cell (DC1) Vaccine; Drug: Trastuzumab; Drug: Pepinemab; Biological: T-Cell therapy
- T-Cell therapy dose level 2 (Experimental): Participants will begin treatment with pepinemab and trastuzumab, and begin DC1 vaccines. After 6 weeks of DC1 vaccines, blood will be collected for t-cell therapy, and patients will then be treated with IL-15 Expanded HER2 specific CD4+ Th1 cell .25-1.2 x 10^9, IL-7 and Expanded HER2 specific CD4+ Th1 cell .25-1.2 x 10^9.
  Interventions: Biological: Dendritic Cell (DC1) Vaccine; Drug: Trastuzumab; Drug: Pepinemab; Biological: T-Cell therapy
- T-Cell therapy dose level 3 (Experimental): Participants will begin treatment with pepinemab and trastuzumab, and begin DC1 vaccines. After 6 weeks of DC1 vaccines, blood will be collected for t-cell therapy, and patients will then be treated with IL-15 Expanded HER2 specific CD4+ Th1 cell .5-2.5 x 10^9, IL-7 and Expanded HER2 specific CD4+ Th1 cell .5-2.5 x 10^9.
  Interventions: Biological: Dendritic Cell (DC1) Vaccine; Drug: Trastuzumab; Drug: Pepinemab; Biological: T-Cell therapy
- T Cell therapy dose expansion (Experimental): Participants will begin treatment with pepinemab and trastuzumab, and begin DC1 vaccines. After 6 weeks of DC1 vaccines, blood will be collected for t-cell therapy, and patients will then be treated with CD4 treated t-cells at the maximum tolerated dose determined.
  Interventions: Biological: Dendritic Cell (DC1) Vaccine; Drug: Trastuzumab; Drug: Pepinemab; Biological: T-Cell therapy

INTERVENTIONS:
Biological: Dendritic Cell (DC1) Vaccine — Participants will receive a DC1 vaccine injection at 1.0-2.0 x 10^7 cells, either to groin lymph notes or to tumor if accessible once a week for 3 weeks on days 1, 8 and 15. Participants will receive DC1 vaccine boosters every 3 weeks x 3.
Drug: Trastuzumab — Participants will receive trastuzumab 8 mg/kg by IV week 1, then 6 mg/kg by IV beginning week 4 and continuing every 3 weeks until disease progression or intolerable toxicity.
  Other Names: Herceptin; Trazimera
Drug: Pepinemab — Participants will receive pepinemab 20 mg/kg by IV beginning week 1 and continuing every 3 weeks until disease progression or intolerable toxicity.
Biological: T-Cell therapy — Participants will receive IL-15 expanded CD4 T cells infusion by IV Day 1 at week 8, 2 weeks from last DC1 vaccine, and IL-7 expanded CD4 T cells infusion IV at week 8 day 8.

SUMMARY:
The purpose of this study is to test the safety of Adoptive T-Cell therapy following the Dendritic Cell (DC1) study vaccine given in combination with pepinemab added to standard of care therapy, trastuzumab to help people with HER2 positive breast cancer.

DETAILED DESCRIPTION:
Patients with HER2-positive (HER2+) metastatic breast cancer will be treated with 6 weekly injections of dendritic cell (DC1) vaccines in combination with trastuzumab and pepinemab.

Investigators hypothesize these therapies will elicit CD4+ HER2 specific T cell responses. HER2 specific T cells will be expanded ex vivo which will be infused to patients subsequently following lymphodepletion therapy with cyclophosphamide. Trastuzumab and pepinemab will be given as maintenance in addition to booster DC1 vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically confirmed HER2 positive breast cancer and must be candidates for trastuzumab therapy as per current standard of care. Note: HER2 positive breast cancer is defined by tumor tissue HER2 overexpression and or tumor HER2 amplification per ASCO/CAP criteria.
* Patients will be eligible regardless of ER/PR status which will be determined per 2020 ASCO/CAP guideline and hormonal therapy will be allowed to continue for patients with ER/PR positive disease.
* Must have evaluable disease, defined as at least one lesion that can be accurately measured ≥ 10 mm by standard imaging techniques that can be include but not limited to CT, PET, PET/CT, MRI. Skeletal disease which is measurable by PET/CT or bone scan will also be allowed.
* Must have had disease progression while on trastuzumab for the treatment of HER2+ MBC and received no more than 3 lines of cytotoxic chemotherapy in the setting of metastatic disease.
* ECOG performance status 0 or 1.
* Must have normal organ and marrow function as defined in protocol within 14 days of registration.
* Left ventricular ejection fraction above institutional lower limit of normal (by echocardiogram or MUGA scan)
* Female patients of childbearing potential must agree to use dual methods of contraception and have a negative serum or urine pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose. To be considered of not to be of childbearing potential, postmenopausal women must be amenorrheic for at least 12 months naturally (not in the setting of post chemotherapy) or patients must be surgically sterile.
* Must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.
* Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 14 days prior to beginning protocol therapy.
* Patients may not be receiving any other investigational agents within 14 days or 5 half-lives (whichever is longer) prior to beginning protocol therapy.
* Patients with uncontrolled brain metastases or leptomeningeal disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded.
* Female patients who are pregnant or nursing are not eligible.
* Second invasive malignancy requiring active treatment
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) is not permitted.
* Any known positive test for Hepatitis B or Hepatitis C virus indicating acute or chronic infection is not permitted.
* Patients who have received a live attenuated vaccine ≤30 days of registration are not eligible.
* Patients not able to comply with the treatment schedule and study procedures for any reason are not eligible.
* Patients previously treated with any form of adoptive cell transfer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of expanded CD4 T cells | Up to 6 months
  MTD of expanded CD4 T cells after treatment with DC1 vaccines and trastuzumab/pepinemab.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 6 months
  ORR according to RECIST criteria v1.1 and iRECIST of treatment DC1 vaccines and pepinemab/trastuzumab
Clinical Benefit Rate (CBR) of DC1 vaccines and pepinemab/trastuzumab | at 6 months
  To assess the 6-month clinical benefit rate (CBR) according to RECIST criteria v. 1.1 of treatment with DC1 vaccines and pepinemab/trastuzumab
Clinical Benefit Rate (CBR) of expanded CD4 T Cells | at 6 months
  To assess the 6-month CBR according to RECIST criteria v. 1.1 of treatment with expanded CD4+ T cells following DC1 vaccines and pepinemab/trastuzumab.
Progression Free Survival (PFS) | Up to 36 months
  PFS is defined as the length of time from start of treatment to progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Han, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No